CLINICAL TRIAL: NCT06509243
Title: Dupilumab and House Dust Mite Immunotherapy in Patients With Atopic Dermatitis
Acronym: DuHDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KNW-1-131/N/9/K
Record Dates: First submitted 2024-06-05; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; biologics; allergen immunotherapy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; Cyclosporine

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled, double-blind 12-month trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SLIT HDM (Active Comparator): Patients received sublingual allergen immunotherapy (Acarizax), adding to symptomatic therapy for atopic dermatitis (according to recommendations).
  Interventions: Biological: tablets Acarizax
- biologic (Active Comparator): Patients received dupilumab, added to symptomatic therapy for atopic dermatitis (according to recommendations.)
  Interventions: Biological: dupilumab
- Combi therapy (Active Comparator): Patients received sublingual allergen immunotherapy (Acarizax) and dupilumab, added to symptomatic therapy for atopic dermatitis (according to recommendations).
  Interventions: Biological: tablets Acarizax; Biological: dupilumab
- cyclosporine (Placebo Comparator): Patients received cyclosporine added to symptomatic therapy for atopic dermatitis (according to recommendations).
  Interventions: Drug: cyclosporine

INTERVENTIONS:
Biological: tablets Acarizax — sublingual immunotherapy to house dust mites
  Arms: Combi therapy; SLIT HDM
Biological: dupilumab — dupilumab - biologic therapy for atopic dermatitis
  Arms: Combi therapy; biologic
Drug: cyclosporine — cyclosporine used in atopic dermatitis
  Arms: cyclosporine

SUMMARY:
Severe atopic dermatitis (AD) is a complex disease requiring systemic treatment. This study aimed to assess the effectiveness of combined therapy consisting of dupilumab and sublingual dust mite allergen immunotherapy (SLIT-HDM) in patients with severe AD and HDM allergies.

Methods: Patients diagnosed with severe AD were included in a randomized, placebo-controlled, double-blind 12-month trial; they received SLIT to HDM and/or dupilumab for 12 months and were compared to patients on cyclosporine. EASI, %BSA, and IsGA changes were analyzed in the different treatment arms from the beginning to the end of the 12th month. The secondary outcomes were the proportion of patients who achieved IsGA success and reduced medication scores.

DETAILED DESCRIPTION:
Study design This randomized, 12-month trial has performed in the Clinical Outpatient Allergy Department and six other outpatient cities. All included patients has received SLIT to HDM and/or dupilumab for 12 months and were compared to patients on cyclosporine.

Patients Patients were eligible if they met the following criteria: were diagnosed with AD a minimum of one year before the study (documented one year of therapy for AD); were between 18 and 45 years of age; had severe AD with an Eczema Area and Severity Index (EASI) >20 points, a %BSA (body surface area) >10 points, an IsGA (Investigator Global Assessment) = 4 points, a positive skin prick test (SPT) and a positive result for specific immunoglobulin E (sIgE) to extracts of D. pteronyssinus and D. farinae and to Der p 1; had negative results for SPT and sIgE to other inhalant allergens; and had no symptoms of allergic asthma and/or allergic rhinitis. The diagnosis of severe AD was based on the guidelines of the Polish Dermatological Society with more restrictive cut-off points on the EASI, %BSA, and IsGA scales, as presented in the inclusion criteria, to limit the study group to the most advanced forms of AD.14

The exclusion criteria included the following: other active dermatoses, systemic immunosuppressant treatment up to 7 months before the study, other chronic diseases, contraindications to sublingual immunotherapy or sarilumab, and lack of written consent. The dermatologist assessed signs of AD at each study visit.

Treatment The patients have received SLIT-HDM (ACARIZAX, ALk Abello, Denmark) with 12 SQ-HDMs of a standardized allergen extract of the house dust mites Dermatophagoides pteronyssinus and Dermatophagoides farinae (50/50%). The Acarizax tablets were removed from the blister unit immediately after opening the blister and placed under the tongue, where they were dissolved. Swallowing was avoided for approximately 2 minutes. Food and beverages were not ingested for 5 minutes after intake of the tablet. The daily dose was one tablet every day for 12 months. Dupilumab treatment was administered according to established recommendations. Briefly, the patient received a single initial dose of 600 mg of dupilumab followed by subsequent doses of 300 mg every 2 weeks.

All patients used emollients. During therapy, patients with clinical signs of bacterially infected skin were allowed to receive treatment with topical mupirocin or/and a 7-day course of amoxicillin or/and prednisolone (0.5 mg/kg) for seven days for any occurrence of skin exacerbation, including superinfection. In the control group, cyclosporine was administered at 3.5 mg/kg at the start of therapy, with the possibility of modifying the dose according to symptoms after a minimum of 6 months of therapy. Further treatment was administered for a minimum of another six months (12 months in total). Treatment was discontinued if adverse effects occurred.

In all groups, oral antihistamines such as desloratadine and topical medications were added depending on the individual disease. If there was clinical worsening of AD (reported significant severity of itching, the appearance of erythroderma, and new skin lesions of a large area), the patient also received oral glucocorticosteroids at a dose of 10 mg of encortolon per 7 days.

Symptomatic treatment was assessed via the following medication scores: one point for daily use of desloratadine, mometasone furoate cream, or mupirocin ointment, 7 points for every course of amoxicillin and 10 points for the course of encortolon. The patients were required to record symptomatic drug use on the diary card

The statistical analysis was performed using Statistica version 8.12 (SoftPol, Cracow, Poland). Nonparametric tests were used because the data were not normally distributed. The Wilcoxon test was used to analyse differences between the groups. ANOVA was used to compare the scale scores. Differences were considered significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with AD a minimum of one year before the study (documented one year of therapy for AD)
* between 18 and 45 years of age
* severe AD with an Eczema Area and Severity Index (EASI) >20 points, a %BSA (body surface area) >10 points, an IsGA (Investigator Global Assessment) = 4 points, a positive skin prick test (SPT)
* a positive result for specific immunoglobulin E (sIgE) to extracts of D. pteronyssinus and D. farinae and to Der p 1;
* negative results for SPT and sIgE to other inhalant allergens;
* no symptoms of allergic asthma and/or allergic rhinitis

Exclusion Criteria:

* other active dermatoses, systemic immunosuppressant treatment up to 7 months before the study, other chronic diseases,
* contraindications to sublingual immunotherapy or dupilumab,
* lack of written consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Changes in EASI (the Eczema Area and Severity Index) scale | 12 months
  objective improvement of skin lesions in the course of atopic dermatitis based on assessment using standardized questionnaire tests EASI. The EASI assessed disease extent on a scale of 0 to 6 in 4 defined body regions plus an assessment of erythema, infiltration, and/or population; excoriation; and lichenification, each on a scale of 0 to 3. A formula was then used to calculate the total score for each of the 4 regions, which were then added together. Interpretation of the EASI result: 0 = no change, 0.1-1.0 = almost no change, 1.1-7.0 = mild in intensity, 7.1-21.0 = moderate intensity, 21.1-50.0 = high intensity, 50.1-72.0 = very severe (points)
Changes in BSA% (Body Surface Area) scale | 12 months
  Ii atopic dermatitis, %BSA was categorised according to severity bands: clear (0%), mild (> 0 to < 16%), moderate (16 to < 40%), and severe (40-100%) (percentage)
Changes in IsGA (investigator global assessment) scale | 12 months
  The IsGA is a doctor-assessed outcome that evaluates overall AD severity on a 5-point scale ranging from clear (0) to severe (4) or very severe (5).

SECONDARY OUTCOMES:
Significant reduction in IsGA scale | 12 months
  the proportion of patients who achieved IsGA success (defined as a ≥2-grade improvement in IsGA from baseline
changes in DLQI (Dermatology Life Quality Index ) questionnaire | 12 months
  DLQI is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. It is de-signed for people aged 16 years and above.
exacerbations of atopic dermatitis | 12 months
  number of exacerbations of atopic dermatitis per year of observation. Definition:in terms of the need to use systemic steroids.
changes in serum concentration of IgG4 against D. pteronyssinus | 12 months
  assessment of allergen-specific IgG4 concentration in blood serum after 6 and 12 months of treatment in arms with the addition of sublingual immunotherapy SLIT-HDM (AU/L)
changes in serum concentration of IgE against D. pteronyssinus | 12 months
  assessment of allergen-specific IgE concentration in blood serum after 6 and 12 months of treatment in arms with the addition of sublingual immunotherapy SLIT-HDM (kU/L)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Bozek, Prof, Principal Investigator — Medical University of Silesia
Locations (1):
- SUM, Zabrze, Poland

REFERENCES:
- [Background] Bogacz-Piaseczynska A, Bozek A. The Effectiveness of Allergen Immunotherapy in Adult Patients with Atopic Dermatitis Allergic to House Dust Mites. Medicina (Kaunas). 2022 Dec 21;59(1):15. doi: 10.3390/medicina59010015. PMID 36676639